CLINICAL TRIAL: NCT07337746
Title: The Effect of Acapella and Incentive Spirometry on Blood Gases and Peak Expiratory Flow Rate After Coronary Artery Bypass Graft: A Randomized Controlled Trial
Brief Title: The Effect of Acapella and Incentive Spirometry on Blood Gases and Peak Expiratory Flow Rate After Coronary Artery Bypass Graft.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Bassima Amir Naji Omar Hilmi, Lecturer, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acapella Device
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Post Opeative Pulmonary Complication
Keywords: Spirometry; Acapella; peak Expiratory Flow Rate; Arterial Blood Gases

STUDY DESIGN:
Intervention Model Description: The study design in the present study was a randomized controlled trial (RCT) design was used in this study to investigate the effect of Acapella and Incentive Spirometry on Blood Gases and Peak Expiratory Flow Rate after Coronary Artery Bypass Graft: A Randomized Controlled Trial. RCT is a quantitative, true experimental, and comparative study executed under controlled conditions, in which interventions are randomly allocated to different groups in order to minimize bias and determine a cause-effect relationship between an intervention and an outcome.
  the population was patients from two cardiac centers selected based on eligibility criteria the. This was achieved through a simple random sampling probability method using two cards. The white card represents the participant included in the study group, and the black card represents patients control the study sample. This method provides researchers with the opportunity to select participants for the study randomly and without bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acapella (oscilatory PEP) (Experimental): Experimental group will take Acapella for 10-15 minutes per session, two times per a day for 2 days before surgery and 3 days after CABG operation.
  Interventions: Device: Acapella therapy
- Incentive Spirometry (Experimental): Experimental group will not be exposed to Acapella and take only Incentive Spirometry for 10-15 minutes per session, 2 times per a day for 2 days before surgery and three consecutive days after CABG Surgery.
  Interventions: Device: Incentive Spirometry therapy
- Routin Care (No Intervention): control group will not be exposed to Acapella or Incentive Spirometry and will take only routine care like breathing exercise, huffing, coughing and manual percussion

INTERVENTIONS:
Device: Incentive Spirometry therapy — is a device that computes the amount of air that is inspired into the lungs. By causing a piston inside the device to raise when breathing in, an incentive spirometer measures the volume of inspired air.
  Arms: Incentive Spirometry
Device: Acapella therapy — Acapella is a vibration-driven respiratory therapy device that breaks up mucus and promotes airway secretions.
  Arms: Acapella (oscilatory PEP)

SUMMARY:
The goal of this clinical trial is to learn if whether the Acapella and Incentive Spirometry have effect on Blood Gas and Peak Expiratory Flow Rate among patients undergoing Coronary Artery Bypass Graft Surgery. the main question it aims to answer is:

* What is the most effect of using a capella versus incentive spirometry on blood gas parameters (pao2 and paco2) and Peak Expiratory Flow Rate in patient undergoing coronary artery bypass grafting?
* is the incentive spirometry have effect on blood gases parameters and Peak Expiratory Flow Rate?
* is the Acapella have effect on blood gas parameters and Peak Expiratory Flow Rate? Researcher will Compare the Level of Blood gases and Peak Expiratory Flow Rate between Coronary Artery Bypass Graft patients who receive Acapella and Incentive Spirometry and those who do not receive it to see if the Acapella and the Incentive Spirometry work to enhance the level of blood gases parameters and Peak Expiratory Flow Rate.

participant will take Acapella and incentive Spirometry on day before surgery and for three days after Surgery for 10-15 min for each session two times a day.

DETAILED DESCRIPTION:
Heart disease has now been eclipsed by cardiovascular diseases as India's leading cause of mortality. The estimated worldwide disease burden surpasses the global average of 235 deaths per 100,000 people, with age-standardized CVD mortality rates of 272 per 100,000. The prevalence of coronary artery disease is on the rise throughout Southeast Asia, with India leading the way in recent years.

CABG is the median sternotomy is the method most frequently used to accomplish it. The process known as "grafting" involves taking a vein or internal mammary artery 3 and placing it both close to and far from the lesion.

The most vulnerable time following surgery is the early postoperative period. The reduction in lung function continues for several months following surgery.

In order to prevent or reduce complications including pneumonia, atelectasis, pulmonary insufficiency, sputum collection, and decreased gas exchange, chest physical therapy has traditionally been a basic part of postoperative care.

Patients undergoing CABG are commonly advised to perform breathing exercises, either with or without mechanical devices, in order to prevent or minimize lung deterioration. A variety of chest physiotherapy techniques are available. These include cough support, early mobilization, posture, incentive spirometry (IS), deep breathing exercises, respiratory muscles, and active cycle breathing techniques (ACBT).

Acapella is a vibration-driven respiratory therapy device that breaks up mucus and promotes airway secretions. It is another method that is frequently utilized. The apparatus can be utilized in any orientation, whether sitting, standing, or lying down, contingent upon the patient's breathing gravity. Acapella Selection is useful. People with lung disease and issues with their excretory system have wide airways. Easily disassembled for improvement, this device is a tremendous asset. The frequency and real resistance of this sludge remover can also be adjusted. In less than half of a natural chest physiotherapy session, patients' management times can also be completed. The Acapella device does not need to be removed by patients while they are using it.

In a variety of clinical contexts, there have been numerous papers demonstrating the benefits of alternate vibration and oscillation on lung function and air outflow. Acapella is made out of a metal bar attached to a handle and magnet, as well as an anti-weight cover. The cause of the oscillation in airflow is the occasional cessation of airflow through the plug, which breaks and repairs the magnetic attraction.

The goal of incentive spirometry is to get the patient to inhale fully, simulate unrestricted yawning or groaning, increase or maintain lung volume, and facilitate the ejection of phlegm.

As a result, the usage of practical tools to facilitate secretory discharge is increasing. Different technologies that support current physiotherapy approaches in increasing mobilization and secretory release have emerged in recent years. Written report focusing on the effectiveness of Acapella as a tool to help with secretion clearance in various lung diseases.

The adverse effects of general anesthesia, intubation, and analgesia on mucociliary clearance following surgery are well documented. When lung volumes are reduced, as they are during the postoperative period, coughing will be less effective since expiratory flow rate is directly correlated with lung volume.

In order to maintain postoperative CABG status, respiratory physiotherapy is essential. Physiotherapists utilize interventions such early mobilization, effective coughing techniques, postoperative breathing exercises, and inspiratory muscle training to promote oxygenation following open heart surgery and minimize lung volume declines and atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is an adult admitted to the hospital for coronary artery bypass graft surgery after receiving a diagnosis of coronary artery disease.
* Been between 33 years and 60 years old.
* being open to taking part in the research and giving informed permission.

Exclusion Criteria:

* individuals having a body mass index (BMI) between 16 and 28 kg/m2.
* patients who have asthma or COPD.
* patients that need reintubation.
* patients who have history of respiratory tract infection.

Ages: 33 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | as baseline one day before surgery (pre-intervention) and post intervention in three consecutive days after surgery.
  For improvement in expiratory airflow indicating lung function recovery
Arterial Blood Gases (ABG) | as a baseline (pre-intervention) one day before surgery and three consecutive days after surgery and post-intervention.
  we see the change in Arterial Blood Gases value before and after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - Ibn AL-Betar Teaching Hospital, Baghdad
  - Iraqi Center of Heart Disease, Baghdad

IPD SHARING:
Plan to Share IPD: No